CLINICAL TRIAL: NCT01708525
Title: Feasibility Study: Determination of the Effect of Ultherapy® Treatment on the Rate of Collagen Synthesis in Normal Skin
Brief Title: Feasibility Study: Heavy Water Tissue Labeling Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-132
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy® Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa | interventions — Deuterium Oxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy®-treated tissue (Experimental): Heavy water labeled tissue receiving an Ulthera® System Treatment
  Interventions: Device: Ulthera® System Treatment; Other: Heavy Water

INTERVENTIONS:
Device: Ulthera® System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy®
Other: Heavy Water — A tissue labeling model via the consumption of the stable isotope, deuterated water (heavy water). Heavy water consumed over the course of the 6-week study period for a direct kinetic measure of in vivo collagen synthesis. 60 ml (about 12 teaspoons) of heavy water (also called deuterated water or 2H2O), was consumed three times a day for the first five days. Starting on Day 6, two 60 ml doses of heavy water were consumed per day for the remaining 37 days.
  Other Names: Deuterated Water

SUMMARY:
Enrolled subjects undergo tissue labeling to evaluate the rate of collagen synthesis in tissue treated with the Ulthera® System compared to control tissue.

DETAILED DESCRIPTION:
This study is a prospective, single-center, blinded, non-randomized clinical trial. Two subjects who have chosen to have a surgical facelift procedure and agree to drink heavy water for tissue labeling, will be enrolled. Subjects will consume heavy water and collect saliva specimens over the course of the study period, following a specific heavy water labeling protocol. Two weeks after starting the heavy water protocol, subjects will return to the study site to receive one Ultherapy® treatment to the pre-auricular region on one side of the face. The contra-lateral pre-auricular region will serve as a control. Following Ultherapy® treatment, subjects will continue to follow the heavy water protocol for 4 more weeks. Subjects will then return to the study site to undergo resection of the treated and control tissue for analysis during their planned rhytidectomy procedure. Subjects will send in saliva samples on a weekly basis to allow for confirmation that they are drinking the heavy water.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 65 years scheduled for rhytidectomy.
* Subject in good health.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1 and be willing and able to use an acceptable method of birth control.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Significant scarring in areas to be treated.
* Open wounds or lesions in the area to be treated.
* Severe or cystic acne on the area to be treated.
* Presence of a metal stent or implant in the facial area to be treated.
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatments to the submental area within two weeks prior to study participation or during the study.
* Excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area to be treated.
* BMI equal to or greater than 30.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Sasaki, MD, Principal Investigator — Sasaki Advanced Aesthetic Medical Center
Locations (1):
- Sasaki Advanced Aesthetic Medical Center, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultherapy®-Treated Tissue: Heavy water labeled tissue receiving an Ultherapy® Treatment
  Ulthera System® Treatment: Focused ultrasound energy delivered below the surface of the skin
Period: Overall Study
Arm/Group | Ultherapy®-Treated Tissue
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Both study subjects completed two weeks of heavy water tissue labeling then received Ultherapy® treatment to the pre-auricular region on one side of their face. The non-treated pre-auricular region on the contralateral side served as a control. Treated and non-treated tissue was resected at 4 weeks post Ultherapy® for analysis.
Arm/Group | Ultherapy®-Treated Tissue
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 62 [59 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Collagen Synthesis
Description: Resected tissue will be analyzed to determine the rate of collagen synthesis in tissue treated with Ultherapy® compared to non-treated tissue.
Time Frame: 4 weeks post-treatment
Measure: Number; unit: percentage of new collagen synthesized
Groups:
- Untreated Tissue: Heavy water labeled tissue NOT receiving an Ultherapy® Treatment
- Ultherapy®-Treated Tissue: Heavy water labeled tissue receiving an Ultherapy® Treatment
  Ulthera® System Treatment: Focused ultrasound energy delivered below the surface of the skin
Arm/Group | Untreated Tissue | Ultherapy®-Treated Tissue
Number analyzed (Participants) | 2 | 2
percentage of new collagen synthesized
  Subject 1, Type I Collagen | 15.71 | 21.22
  Subject 1, Type III Collagen | 36.11 | 51.80
  Subject 2, Type I Collagen | 18.53 | 29.69
  Subject 2, Type III Collagen | 50.34 | 68.13

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through tissue resection, i.e., 4 weeks post-Ultherapy® treatment.
Arm/Group | Ultherapy®-Treated Tissue
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
A limitation of this trial includes only a two subject study population due to the extremely high expense of the tissue analyses conducted. High expense precluded further research in a randomized designed trial with a broader patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No